CLINICAL TRIAL: NCT00011674
Title: Early Exposure to Lead and Adolescent Development
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Other Study IDs: 8158-CP-001
Record Dates: First submitted 2001-02-26; First posted 2001-02-28 (Estimated); Last update posted 2006-03-23 (Estimated); Status verified 2006-03

CONDITIONS: Lead Poisoning
Keywords: Lead; Prenatal; Development; Children; Psychology; Toxicology; Teratology
MeSH Terms: conditions — Lead Poisoning

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
This prospective cohort study examines the role of prenatal and early postnatal lead exposure on the neuropsychological status and social adjustment of adolescents enrolled in the Cincinnati Lead Study. We are examining the relationship between moderate exposure to lead and neuropsychological deficits, difficulties in peer relationships, personality disturbances and juvenile delinquency. This birth cohort of approximately 300 subjects has been followed since 1980 with regularly scheduled assessments of blood lead concentrations, health history, social and hereditary factors, and neurobehavioral development.

ELIGIBILITY:
Subjects for the Cincinnati Lead Study were recruited prenatally if their mothers resided in areas within Cincinnati, Ohio where there has historically been a high incidence of lead poisoning. Infants were eligible for follow-up if they were greater than 1500 grams at birth and had no disqualifying medical conditions such as defined genetic syndromes or other serious complications that may adversely affect neurobehavioral development.

Min Age: 0 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 300
Dates: Start 1997-05; Study Completion 2001-05

CONTACTS AND LOCATIONS:
Locations (1):
- Findlay Street Clinic, Cincinnati, Ohio, United States